CLINICAL TRIAL: NCT06878391
Title: A Study on the Pain Control Effects of Interscalene Brachial Plexus Block Combined With Suprascapular Nerve Block and Axillary Nerve Block in Ar-throscopic Rotator Cuff Repair: a Randomized Controlled Trial
Brief Title: ISB With SSNB & ANB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Jung-Taek Hwang, Professor, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2024-12-010-003
Record Dates: First submitted 2025-03-13; First posted 2025-03-17 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-03

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Intervention Model Description: Study group: Preemptive US guided interscalene brachial plexus block (9ml 0.75% ropivacaine, 3ml for each trunk), and suprascapular nerve block (SSNB) and axillary nerve block (ANB) using each 0.75% ropivacaine 10mL Control group: Preemptive US guided interscalene brachial plexus block (9ml 0.75% ropivacaine, 3ml for each trunk), and suprascapular nerve block (SSNB) and axillary nerve block (ANB) using each 0.9% saline 10mL
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An independent nurse uses a random number generator and allocates paticipants into the two group. Participant, investigator, and outcome assessor are blinded of the allocation information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ISB with SSNB & ANB (Experimental): An ultrasound-guided interscalene brachial plexus block (9 ml of 0.75% ropivacaine, 3 ml for each trunk) is performed immediately before arthroscopic rotator cuff repair , along with suprascapular nerve block and axillary nerve block (each with 10 ml of 0.75% ropivacaine). Patient Controlled Analgesia (PCA) at a low fixed dose: fentanyl-loading dose: 0.4㎍/kg, continuous dose: 0.2㎍/kg/h, nefopam-loading dose: 0.04mg/kg, continuous dose: 0.02mg/kg/h
  Interventions: Procedure: Preemptive ultrasound-guided interscalene brachial plexus block and suprascapular nerve block and axillary nerve block
- ISB with placebo SSNB & ANB (Placebo Comparator): An ultrasound-guided interscalene brachial plexus block (9 ml of 0.75% ropivacaine, 3 ml for each trunk) is performed immediately before arthroscopic rotator cuff repair , along with suprascapular nerve block and axillary nerve block (each with 10 ml of saline). Patient Controlled Analgesia (PCA) at a low fixed dose: fentanyl-loading dose: 0.4㎍/kg, continuous dose: 0.2㎍/kg/h, nefopam-loading dose: 0.04mg/kg, continuous dose: 0.02mg/kg/h
  Interventions: Procedure: Preemptive ultrasound-guided interscalene brachial plexus block and suprascapular nerve block and axillary nerve block

INTERVENTIONS:
Procedure: Preemptive ultrasound-guided interscalene brachial plexus block and suprascapular nerve block and axillary nerve block — Preemptive ultrasound-guided interscalene brachial plexus block using ropivacaine, and suprascapular nerve block and axillary nerve block using ropivacaine or saline. Low fixed dose patient controlled analgesia (PCA) were done in the two group.
  Other Names: a low fixed dose patient controlled analgesia (PCA)

SUMMARY:
This study is a prospective, randomized, double-blind trial comparing patients who underwent arthroscopic rotator cuff repair and received an interscalene brachial plexus block (9 ml of 0.75% ropivacaine, 3 ml for each trunk) combined with suprascapular nerve block and axillary nerve block (each with 10 ml of 0.75% ropivacaine) versus those who received an interscalene brachial plexus block (9 ml of 0.75% ropivacaine, 3 ml for each trunk) combined with placebo suprascapular and axillary nerve blocks (each with 10 ml of 0.9% saline).

The study will compare subjective pain scores (VAS score) and patient satisfaction preoperatively and at 1, 3, 6, 12, 18, 24, 36, and 48 hours postoperatively. Additionally, 5 ml of venous blood will be collected preoperatively and at 1, 6, 12, 24, and 48 hours postoperatively to analyze and compare serum levels of cortisol, IL-6, IL-8, IL-1β, substance P, serotonin, β-endorphin, and norepinephrine.

ELIGIBILITY:
Inclusion Criteria:

* a definite rotator cuff tear that needed repair seen on preoperative magnetic resonancce imaging (MRI)
* acceptance of arthroscopic surgery including rotator cuff repair
* age same as or more than 20 years
* acceptance of preemptive regional block and PCA, and blood testing

Exclusion Criteria:

* did not undergo arthroscopic rotator cuff repair
* stopped PCA before 48 hours postoperatively because of associated side effects
* a history of previous ipsilateral shoulder operation or fracture
* a concomitant neurologic disorder around the shoulder
* a failure of blood sampling including hemolysis, etc.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
visual analog pain scale (VAS) | preoperative, postoperative 1, 3, 6, 12, 18, 24, 36, 48 hour(s)
  0-10, 0: no pain, 10: very severe pain

SECONDARY OUTCOMES:
Patient's satisfaction (SAT) | preoperative, postoperative 1, 3, 6, 12, 18, 24, 36, 48 hour(s)
  0-10, 0: not satisfied, 10: very much satisfied
plasma Cortisol | preoperative, postoperative 1, 6, 12, 24, 48 hour(s)
  ng/mL
IL-6 | preoperative, postoperative 1, 6, 12, 24, 48 hour(s)
  pg/mL
IL-8 | preoperative, postoperative 1, 6, 12, 24, 48 hour(s)
  pg/mL
IL-1β | preoperative, postoperative 1, 6, 12, 24, 48 hour(s)
  pg/mL
Substance P | preoperative, postoperative 1, 6, 12, 24, 48 hour(s)
  pg/mL
Serotonin | preoperative, postoperative 1, 6, 12, 24, 48 hour(s)
  ng/mL
β -endorphin | preoperative, postoperative 1, 6, 12, 24, 48 hour(s)
  pg/mL
norepinephrine | preoperative, postoperative 1, 6, 12, 24, 48 hour(s)
  pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Taek Hwang, MD, PhD, Principal Investigator — Hallym University Medical Center
Locations (1):
- Hallym University Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No
We can decide it after the termination of this study.

REFERENCES:
- [Background] Lee JJ, Kim DY, Hwang JT, Lee SS, Hwang SM, Kim GH, Jo YG. Effect of ultrasonographically guided axillary nerve block combined with suprascapular nerve block in arthroscopic rotator cuff repair: a randomized controlled trial. Arthroscopy. 2014 Aug;30(8):906-14. doi: 10.1016/j.arthro.2014.03.014. Epub 2014 May 29. PMID 24880194
- [Background] Lee JJ, Kim DY, Hwang JT, Song DK, Lee HN, Jang JS, Lee SS, Hwang SM, Moon SH, Shim JH. Dexmedetomidine combined with suprascapular nerve block and axillary nerve block has a synergistic effect on relieving postoperative pain after arthroscopic rotator cuff repair. Knee Surg Sports Traumatol Arthrosc. 2021 Dec;29(12):4022-4031. doi: 10.1007/s00167-020-06288-8. Epub 2020 Sep 25. PMID 32975624